CLINICAL TRIAL: NCT01152827
Title: Phase II Study of RAD001monotherapy in Patients With Unresectable Pheochromocytoma or Extra-adrenal Paraganglioma or Non-functioning Carcinoid
Brief Title: RAD001 in Pheochromocytoma or Nonfunctioning Carcinoid
Acronym: PheoCarcRAD001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-0710-049-223
Record Dates: First submitted 2010-05-31; First posted 2010-06-29 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2010-06

CONDITIONS: Pheochromocytoma; Extra-adrenal Paraganglioma; Non-functioning Carcinoid
Keywords: Pheochromocytoma; extra-adrenal paraganglioma; non-functioning carcinoid; RAD001
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma, Extra-Adrenal | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): RAD001 10 mg daily po medication
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 10 mg daily po medication.
  Treatments will be continued until any of the following events occur
  * progression of disease
  * the subject develops unacceptable toxicity
  * consent to participate in the study is withdrawn

SUMMARY:
* According to Martin F et al, AKT is highly phosphorylated in phenochromocytoma but not in benign adrenocortical tumors.
* In nonfunctioning carcinoid, the PI3K/AKT/mTOR pathway is activated.
* Although mTOR is clearly an attractive therapeutic target in tumor, no clinical study on mTOR inhibition by RAD001 have been conducted in pheochromocytoma or extra-adrenal paraganglioma or non-functioning carcinoid.
* So we design this phase II study of RAD001 in pheochromocytoma or extra-adrenal paraganglioma or non-functioning carcinoid to evaluate the efficacy of RAD001 in this orphan disease.

DETAILED DESCRIPTION:
Although several therapeutic options exist for patients with metastatic pheochromocytoma, all options are limited and there is no cure. Reduction of tumor size palliates symptoms, but a survival advantage of debulking is unproven. A reduced tumor burden can facilitate subsequent radiotherapy or chemotherapy. External-beam irradiation of bone metastases and radio frequency ablation of lesions are treatment alternatives. Chemotherapy with a combination of cyclophosphamide, vincristin, and dacarbazine can provide tumor regression and symptom relief in up to 50% of patients, but the responses are usually short-lived. To date, 131I-labeled MIBG therapy is the single most valuable adjunct to surgical treatment of malignant pheochromocytomas. As a single agent, 131I-labeled MIBG has a limited efficacy of cure, and there is no consensus on what doses to use for treating either bone or organ metastases. Multicenter studies are required to reach a consensus on the efficacy of high-dose versus fractionated medium doses of 131I-labeled MIBG and monotherapy versus combination therapy with other radio nuclides or modes of chemotherapy.

The PI3-K/Akt/mTOR pathway is dysregulated in many cancers and is activated by several upstream proteins, such as ras, TCL1, and bcr-abl, and membrane receptor tyrosine kinases, including vascular endothelial growth factor receptor, platelet-derived growth factor receptor, c-kit, and Flt3. Increased expression and constitutive activation of the catalytic subunit of PI3-K and Akt and/or decreased or absent PTEN protein expression have been reported in many types of cancer. Activating mutation in PIK3CA, the gene for the catalytic subunit of PI3-K have been reported in 25% of gastric cancer.

Upstream in the growth-promoting pathways that converge on mTOR are critical molecules that are often deregulated in cancer. These deregulated molecules precede inappropriate signals that activate the mTOR switch, driving the growth and proliferation of the cancer cell. Because the number of potential defects that can cause inappropriate activation of mTOR is large and one or another is common to most cancer cells, blocking their effect at the point of convergence is a rational approach.

According to Martin F et al, AKT is highly phosphorylated in phenochromocytoma but not in benign adrenocortical tumors.

Although mTOR is clearly an attractive therapeutic target in tumor, no clinical study on mTOR inhibition by RAD001 have been conducted in pheochromocytoma or extra-adrenal paraganglioma.

So we conduct this phase II study of RAD001 in this disease And we also include the nonfunctioning carcinoid in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed pheochromocytoma or extra-adrenal paraganglioma or carcinoid
* 2. Local, locally-advanced or metastatic disease documented as having shown progression on a scan (CT, MRI, MIBI scan) taken 2 to 12 months prior to baseline compared to a previous scan taken at any time in the past. Progression must be documented according to RECIST criteria.
* 3. Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent.
* 4. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria
* 5. 18 years or older
* 6. ECOG performance status 0, 1
* 7. Previous treatment with chemotherapy, loco-regional therapy (e.g chemoembolization) are permitted providing that toxicity has resolved to ≤grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment.
* 8. Adequate organ function
* 9. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
* 10. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

* 1. A patient with no measurable disease
* 2. Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target lesions (within 2 weeks prior to study entry)
* 3. A patient with functioning carcinoid
* 4. A patient with previous active or passive immunotherapy
* 5. A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding
* 6. A pregnant or lactating patient
* 7. A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential)
* 8. A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study
* 9. A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of skin and cervical carcinoma in situ.
* 10. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
* 11. A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.
* 12. Ongoing cardiac arrhythmia of grade ≥2, atrial fibrillation of any grade, or QTc interval>450msec for males or >470msec for female.
* 13. A patient with interstitial pneumonia or diffuse symptomatic fibrosis of the lungs
* 14. A patient with peripheral neuropathy of grade 1 by NCI CTC, caused by other factors (e.g. alcohol, diabetes, etc). If the absence of deep tendon reflexes is the only neurologic disorder, this condition does not apply to the exclusion criteria.
* 15. A patient with organ transplantation requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
progression-free survival rate at 4 months | 10 months
  proportion of patients who are alive and progression-free at the time of 4 months of treatment among all patients

SECONDARY OUTCOMES:
time to progression (TTP) | 10 months
overall survival (OS) | 2 years
response rate (RR) | 6 months
metabolic response rate by PET-CT | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Jue Bang, MD, PhD, Principal Investigator — Seoul National University Hospital; Do-Youn Oh, MD, PhD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea